CLINICAL TRIAL: NCT02244203
Title: Investigation of Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single Rising Oral Doses of 0.25, 0.5, 1, 2, 4, 20, 50, 100, 150 and 200 mg BI 60732 Powder in Bottle (PIB) Administered to Healthy Male Volunteers in a Randomised, Double Blind, Placebo Controlled Phase I Trial
Brief Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of BI 60732 in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 1267.1
Record Dates: First submitted 2014-09-18; First posted 2014-09-19 (Estimated); Last update posted 2014-09-19 (Estimated); Status verified 2014-09

CONDITIONS: Healthy

ARMS (2):
- Single rising doses of BI 60732 (Experimental)
  Interventions: Drug: BI 60732
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BI 60732
  Arms: Single rising doses of BI 60732
Drug: Placebo
  Arms: Placebo

SUMMARY:
Single Rising Dose (SRD) study: First evaluation of safety, tolerability, pharmacokinetics and pharmacodynamics of BI 60732

ELIGIBILITY:
Inclusion Criteria:

* Healthy males according to the following criteria: Based upon a complete medical history, including the physical examination, vital signs (BP, PR), 12-lead ECG, clinical laboratory tests
* Age ≥ 18 and Age ≤ 45 years
* BMI ≥ 18.5 and BMI ≤ 29.9 kg/m2 (Body Mass Index)
* Signed and dated written informed consent prior to admission to the study in accordance with good clinical practice and the local legislation

Exclusion Criteria:

* Any finding of the medical examination deviating from normal and of clinical relevance. Repeated measurement of a systolic blood pressure greater than 140 mm Hg or diastolic blood pressure greater than 90 mm Hg
* Any evidence of a clinically relevant concomitant disease
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Surgery of the gastrointestinal tract (except appendectomy)
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* History of relevant orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of relevant allergy/hypersensitivity (including allergy to drug or its excipients)
* Intake of drugs within one month or less than 10 half-lives of the respective drug prior to first study drug administration except if a relevant interaction can be ruled out
* Participation in another trial with an investigational drug within 2 months prior to first study drug administration
* Smoker (> 10 cigarettes or > 3 cigars or > 3 pipes/day)
* Alcohol abuse (average consumption of more than 30 g / day)
* Drug abuse
* Blood donation (more than 100 mL within four weeks prior to the start of study)
* Any laboratory value outside the reference range that is of clinical relevance
* Inability to comply with dietary regimen of trial site
* A marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval >450 ms)
* A history of additional risk factors for Torsade de pointes (e.g., heart failure, hypokalaemia, family history of Long QT Syndrome)
* Anaemia at screening
* Subjects who in the investigator's judgement are perceived as having an increased risk of bleeding, for example because of:

  * Hemorrhagic disorders or bleeding diathesis
  * Occult blood in faeces or haematuria
  * Trauma or surgery within the last month or as long as an excessive risk of bleeding persists after these events, or planned surgery during trial participation
  * History of arteriovenous malformation or aneurysm
  * History of gastroduodenal ulcer disease or gastrointestinal haemorrhage
  * History of intracranial, intraocular, spinal, retroperitoneal, or atraumatic intraarticular bleeding
  * Use of drugs that may interfere with haemostasis during trial conduct (e.g. acetylsalicylic acid or other non-steroidal anti-inflammatory drugs)
  * Thrombocytopenia (platelet count < 100/nL)

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2009-02; Primary Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Number of patients with clinically relevant changes in vital signs (blood pressure (BP), pulse rate (PR)) | up to day 21 after start of treatment
Number of patients with clinically relevant changes in 12-lead ECG | up to day 21 after start of treatment
Number of patients with clinically relevant changes in laboratory parameters | up to day 21 after start of treatment
Number of patients with clinically relevant changes in coagulation parameters | up to 72 hours after start of treatment
  Parameters:
  * Activated partial thromboplastin time (aPTT)
  * Prothrombin time (PT)
  * HepTest®
Number of patients with adverse events | up to 6 weeks
Global assessment of tolerability by investigator on a 4-point scale | up to 21 days after start of treatment

SECONDARY OUTCOMES:
Maximum measured concentration of the analyte in plasma (Cmax) | up to 264 hours after start of treatment
Time from dosing to maximum measured concentration of the analyte in plasma (tmax) | up to 264 hours after start of treatment
Area under the concentration-time curve of the analyte in plasma (AUC) | up to 264 hours after start of treatment
Terminal rate constant of the analyte in plasma (λz) | up to 264 hours after start of treatment
Terminal half-life of the analyte in plasma (t1/2) | up to 264 hours after start of treatment
Mean residence time of the analyte in the body after oral administration (MRTpo) | up to 264 hours after start of treatment
Apparent clearance of the analyte in plasma after extravascular administration (CL/F) | up to 264 hours after start of treatment
Amount of analyte eliminated in urine from the time point t1 to time point t2 (Aet1-t2) | up to 264 hours after start of treatment
Fraction of analyte eliminated in urine from time point t1 to time point t2 (fet1-t2) | up to 264 hours after start of treatment
Renal clearance of the analyte from the time point t1 until the time point t2 (CLR,t1-t2) | Pre-dose, up to 264 hours after start of treatment
Changes in activated partial thromboplastin time (aPTT) | Pre-dose, up to 72 hours after start of treatment
Changes in prothrombin time (PT) | Pre-dose, up to 72 hours after start of treatment
Prolongation of coagulation time by Heptest® | up to 72 hours after start of treatment
Inhibition of FXa activity | Pre-dose up to 168 hours after start of treatment
  Russel's Viper Venom (RVV)
Percentage inhibition of endogenous thrombin generation | up to 24 hours after start of treatment
Percentage peak inhibition of thrombin generation | up to 24 hours after start of treatment
Relative prolongation of time to maximum inhibition of thrombin generation | up to 24 hours after start of treatment
Relative prolongation of lag time of thrombin generation | up to 24 hours after start of treatment
Maximum effect (Emax) | up to 168 hours after start of treatment
Time to maximum effect (tmax) | up to 168 hours after start of treatment
Area under the effect curve (AUEC) | up to 168 hours after start of treatment